CLINICAL TRIAL: NCT02609945
Title: A Phase 1 First in Human Open-Label Study of the Safety and Pharmacokinetics of Single Ascending Doses of CVT-427 (Zolmitriptan Inhalation Powder) In Healthy Adults
Brief Title: Safety and Pharmacokinetics (PK) Study of Single Ascending Doses of CVT-427 (Zolmitriptan Inhalation Powder) In Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Acorda Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TRIP-AM-1035
Record Dates: First submitted 2015-11-16; First posted 2015-11-20 (Estimated); Last update posted 2016-06-06 (Estimated); Status verified 2016-06

CONDITIONS: Migraine
Keywords: Migraine attacks
MeSH Terms: conditions — Migraine Disorders | interventions — zolmitriptan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CVT-427 (zolmitriptan inhalation powder) (Experimental): Periods 1-2: Subjects will receive Zomig oral tablet in Period 1 and Zomig nasal spray in Period 2, 1 hour apart.
  Periods 3-6: Subjects will receive CVT-427 (dose levels (DL) 1, 2, 3 and 4), administered in ascending order provided that safety and tolerability data are observed to be adequate to allow dose escalation, approximately 24 hours after preceding DL.
  Interventions: Drug: zolmitriptan; Drug: CVT-427 (zolmitriptan inhalation powder),

INTERVENTIONS:
Drug: zolmitriptan — Oral Tablet and Nasal Spray
  Other Names: Zomig®
Drug: CVT-427 (zolmitriptan inhalation powder), — Capsules containing zolmitriptan; dose levels equivalent to estimated fine particle dose (i.e., lung-delivered) zolmitriptan.

SUMMARY:
This study is the first study in humans with CVT-427 (zolmitriptan inhalation powder) and is designed to evaluate the safety, tolerability, and PK of single ascending doses of CVT-427 in adult healthy volunteers.

DETAILED DESCRIPTION:
Objectives:

* To evaluate the overall safety and tolerability of single, inhaled doses of CVT-427 (zolmitriptan inhalation powder) in healthy adults, with special emphasis on cardiopulmonary effects.
* To describe the pharmacokinetics (PK) of single, inhaled doses of CVT-427, Zomig® Tablet, and Zomig® Nasal Spray in healthy adults.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult men or women volunteers aged 18 to 65 years, inclusive;
* Triptan-naïve;
* Body mass index (BMI) between 18 to 30 kg/m2;
* Forced expiratory volume in one second (FEV1) greater than 80% of predicted for race, age, sex, and height and FEV1/FVC (forced vital capacity) ratio greater than or equal to 70%;
* No history of asthma;
* Non-smoking for at least 5 years;
* In good general health with no clinically significant abnormalities or recognized cardiovascular risk factors that preclude use of triptans and that would interfere with participation in this study as determined by medical history, physical examination, electrocardiogram, and clinical laboratory test results; and negative tests for drug and alcohol, serology, and for pregnancy for female subjects of childbearing potential.

Exclusion Criteria:

* Subject who is not surgically sterile or female subject who is less than 2 years postmenopausal, and who does not agree to use a highly effective birth control method during the study and up to 3 months after the last dose of investigational product;
* Any cardiovascular risk factor including clinically relevant ECG parameter (e.g., PR interval, QRS deviation) or other clinically significant ECG abnormality;
* History of asthma (including exercise-induced asthma and cold-induced asthma) or chronic obstructive pulmonary disorder (COPD) requiring intermittent or continuous use of any oral or inhaled medication therapy within last 3 years;
* Any flu-like syndrome or other respiratory infections within 4 weeks of CVT-427 administration;
* Unable to tolerate blood draws.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2015-11; Primary Completion 2015-12 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Number of patients with adverse events (AEs) including serious AEs | up to 23 days
Pulmonary function | within 90 min prior to dosing and at specified time points up to 24 hours post-dose
  Measured by spirometry using the guideline specified by the Third National Health and Nutrition Examination Survey (NHANES III)
Maximum observed plasma drug concentration (Cmax) | within 15 minutes pre-dose and at specified time points up to 24 hours post-dose
Time to maximum observed plasma drug concentration (Tmax) | within 15 minutes pre-dose and at specified time points up to 24 hours post-dose
Area under the concentration time curve (AUC) | within 15 minutes pre-dose and at specified time points up to 24 hours post-dose
Terminal elimination half-life (t½) | within 15 minutes pre-dose and at specified time points up to 24 hours post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Eisen, MD, Study Director — Acorda Therapeutics
Locations (2):
- United States (2):
  - Site 001, Daytona Beach, Florida
  - Site 002, Dallas, Texas